CLINICAL TRIAL: NCT06418828
Title: Cross-sectional Survey and Prediction Model Construction of Patients With Type B Aortic Dissection Returning to Work After Discharge
Brief Title: Patients With Type B Aortic Dissection Returning to Work After Discharge：a Cross-sectional Survey
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024KY049
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Type B Aortic Dissection; Return to Work
MeSH Terms: interventions — Return to Work

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Return to work group: Asked whether the patient returned to work, if the patient returned to work, included in this group.
  Interventions: Other: return to work
- Non-return to work group: Ask whether the patient returned to work, if the patient did not return to work, included in this group.
  Interventions: Other: return to work

INTERVENTIONS:
Other: return to work — Ask patients if they are going back to work

SUMMARY:
This study wants to understand the incidence of returning to work after discharge in patients with type B aortic dissection.

DETAILED DESCRIPTION:
The incidence of aortic dissection in China is increasing year by year. According to the latest research report, the annual incidence of aortic dissection in China is 5 ~ 10 / 100,000, the average age of patients is 51.8 years old, and the age of disease is about 10 years younger than that of European and American countries. RTW after discharge is a measure of disease recovery and recovery to normal state. There are only reports on RTW after discharge in the fields of cancer, stroke, organ transplantation, maintenance peritoneal dialysis and so on. Most of the existing literature in the cardiovascular field at home and abroad focuses on assessing the status of RTW and RRTW after discharge. Up to now, there is still a lack of research on the promotion and hindrance factors of RTW in TBAD patients, the status survey of post-RTW work ability and the related nomogram prediction model. Therefore, based on the Meleis transformation theory, this study aims to investigate the current status of return to work of TBAD patients at 6 months after discharge through quantitative and qualitative research, and to explore its influencing factors in depth. Based on the previous results, the RTW visual prediction model of TBAD patients was constructed, which provided a theoretical basis for the formulation and implementation of early intervention by medical staff, and further improved the research in this field.

ELIGIBILITY:
Inclusion Criteria:

( 1 ) TBAD was diagnosed by computed tomography angiography ( CTA ) or magnetic resonance angiography ( MRA ) ; ( 2 ) 18 years ≤ age < 60 years at diagnosis ; ( 3 ) having full-time or part-time job at the time of diagnosis ; ( 4 ) TBAD patients were discharged after successful treatment and the discharge time was ≥ 6 months ;

Exclusion Criteria:

( 1 ) reaching the retirement age 6 months after discharge ; ( 2 ) those with disturbance of consciousness, mental illness, inability to complete the interview independently or under the guidance of the researcher ; ( 3 ) Participate in other related research ; ( 4 ) Clinical end-stage or receiving palliative treatment.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: This study selected patients with TBAD who were hospitalized in the Department of Cardiac Surgery, Union Hospital Affiliated to Fujian Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of return to work | Six months after discharge,
  the incidence of returning to work was calculated according to whether the included patients could return to work.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No